CLINICAL TRIAL: NCT02409901
Title: Randomized Case-Control Trial About the Impact of Targeted Physical Activity and Diet Modification on Kidney Transplant Recipients' Outcome
Brief Title: Effects of Personalized Physical Rehabilitation in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Enrico Benedetti, Professor and Head of Department of Surgery, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-0808
Record Dates: First submitted 2015-03-26; First posted 2015-04-07 (Estimated); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Kidney Transplant
Keywords: Physical Activity; Exercise Rehabilitation; Kidney Function; Employment; Kidney Transplant
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Rehabilitation (Experimental): 12 month personalized exercise rehabilitation in addition to standard clinical care
  Interventions: Behavioral: Exercise Rehabilitation
- Control (No Intervention): Standard clinical care only

INTERVENTIONS:
Behavioral: Exercise Rehabilitation — 12 month personalized exercise rehabilitation in addition to standard clinical care
  Arms: Exercise Rehabilitation

SUMMARY:
This randomized controlled trial (RCT) will examine the effect of a novel 12 month personalized exercise rehabilitation program compared to standard care following kidney transplantation. Return to work or find work rates, markers of subclinical atherosclerosis, functional capacity, body composition, quality of life, kidney function, and adherence to exercise will be measured. The investigators' primary hypothesis is that a 12 month exercise rehabilitation program will increase the return to work or find work rate in kidney transplant recipients. The investigators additionally hypothesize that a 12 month exercise rehabilitation program will prevent a decline in subclinical atherosclerosis, increase functional capacity, and increase lean muscle mass.

DETAILED DESCRIPTION:
The proposed study, data collection, and intervention will be performed in the Integrative Physiology Laboratory at the University of Illinois at Chicago. Blood samples will be collected in the Transplant Clinic at the University of Illinois at Chicago. The study will use a two-arm RCT design to examine the effects of personalized exercise rehabilitation versus standard clinical care in kidney transplant (KT) recipients. The primary outcome will be patient return to work/find work rates. Secondary outcomes will include physical and vascular function, body composition, perceived quality of life, kidney function and blood lipid markers, and adherence. 120 kidney transplant recipients will be randomized 2:1 into either an exercise rehabilitation program or a control group, which involves standard clinical care only. Randomization will be done after obtaining informed consent and baseline testing, utilizing a computerized randomization program as a way to prevent potential selection bias. The exercise rehabilitation arm includes low intensity, personalized resistance trainings two times per week for a 12 month period in addition to standard clinical care (including regular check-ups and blood work as recommended by their post-transplant physician). The control group will continue standard care as advised by their post-transplant medical team with no additional intervention. The investigator will collect data on employment status, and all physiological and psychological data at baseline (before intervention), during (6 months), and immediately after the intervention (12 months). Adherence will be monitored throughout the entirety of the study by recording study visits as well as having the exercise trainers keep record of the patient's attendance in the exercise arm. A 2 X 3 (condition X time) mixed factor, analysis of variance with intent-to-treat principles will be utilized for testing the effect of the intervention on the outcome variables. The investigators' primary hypothesis is that a 12 month exercise rehabilitation program will increase the return to work/find work rate in kidney transplant recipients. It is additionally hypothesize that a 12 month exercise rehabilitation program will prevent a decline in subclinical atherosclerosis, increase functional capacity, and increase lean muscle mass. Outcome measures for subclinical atherosclerosis include aortic pulse wave velocity (PWV), carotid intima-media thickness (IMT), endothelial function and carotid arterial stiffness. The outcome measures for functional capacity include the 6 minute walk test (6MW), unilateral isometric strength test, and free-living accelerometry. Fat and lean muscle mass will be assessed via Dual-energy X-ray absorptiometry (DXA). Quality of life and perceptions of pain will be assessed utilizing the Patient Reported Outcomes Measurement Information System (PROMIS) Global health and PROMIS 29 v 2 questionnaires. Additionally, fasting blood lipid profile, inflammatory markers, and markers of kidney function including glomerular filtration rate (GFR) and creatinine levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 moths post-transplant
* must have adequate cognitive ability to complete questionnaires, give consent for the study and follow the physical instructions

Exclusion Criteria:

* any other organ besides kidney or kidney/pancreas mix
* any surgery or procedure to assist in weight loss (ie bariatric surgery)
* non-ambulatory or significant orthopedic problems
* cardiac/pulmonary disease that contraindicates the physical training
* any contraindication to exercise testing per the American Heart Association
* if the patient is unable to comply with the training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-10; Primary Completion 2019-04 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kastelz A, Fernhall B, Wang E, Tzvetanov I, Spaggiari M, Shetty A, Gallon L, Hachaj G, Kaplan B, Benedetti E. Personalized physical rehabilitation program and employment in kidney transplant recipients: a randomized trial. Transpl Int. 2021 Jun;34(6):1083-1092. doi: 10.1111/tri.13868. Epub 2021 Apr 11. PMID 33733479

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Rehabiliation: 12 month personalized exercise rehabilitation in addition to standard clinical care
  Exercise Rehabilitation: 12 month personalized exercise rehabilitation twice a week, in addition to standard clinical care
Period: Overall Study
Arm/Group | Exercise Rehabiliation | Control
Started | 93 | 42
Completed Baseline Assessment (Those number of patients have baseline characteristics collected) | 80 | 33
Completed (Completed data analysis) | 52 | 28
Not Completed | 41 | 14

BASELINE CHARACTERISTICS:
Groups:
- Exercise Rehabiliation: 12 month personalized exercise rehabilitation in addition to standard clinical care
  Exercise Rehabilitation: 12 month personalized exercise rehabilitation in addition to standard clinical care
- Total: Total of all reporting groups
Arm/Group | Exercise Rehabiliation | Control | Total
Number analyzed (Participants) | 80 | 33 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.29 (11.56) | 43.18 (11.98) | 45.24 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 48 | 15 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 54 | 21 | 75
  White | 10 | 2 | 12
  More than one race | 13 | 10 | 23
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 80 | 33 | 113

OUTCOME MEASURES:

1. Primary Outcome: Employment Status
Description: This will be assessed through verbal questioning on the current employment status of each participant.
  Overall number of participants only includes participants who were unemployed at baseline.
Time Frame: 12 months
Population: The count represents the number of participants who were unemployed at Baseline (excluding employed participants at baseline)
Measure: Count of Participants; unit: Participants
Groups:
- Exercise Rehabilitation: 12 month personalized exercise rehabilitation in addition to standard clinical care
  Exercise Rehabilitation: 12 month personalized exercise rehabilitation twice a week, in addition to standard clinical care
Arm/Group | Exercise Rehabilitation | Control
Number analyzed (Participants) | 44 | 15
Participants | 21 | 2

2. Secondary Outcome: Subclinical Atherosclerosis - PWV
Description: This will be assessed through measures of aortic pulse wave velocity (PWV)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
meters/second | 7.16 (2.31) | 6.06 (1.96)

3. Secondary Outcome: Functional Capacity - 6MW
Description: This will be assessed through the 6 minute walk test (6MW). The test measures the distance (in meters) patients can walk in 6 minutes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
Meters | 418.41 (111.65) | 405.95 (95.79)

4. Secondary Outcome: Body Composition - DEXA
Description: Muscle mass will be assessed via Dual-energy X-ray absorptiometry (DEXA).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Gram
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
Gram | 2858.10 (678.12) | 2550.69 (431.37)

5. Secondary Outcome: Metabolic State and Kidney Function - eGFR
Description: Estimated glomerular filtration rate (eGFR) will be measured
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
mL/min/1.73m^2 | 57.46 (20.91) | 62.48 (17.70)

6. Secondary Outcome: Quality of Life and Perceived Health Status - PROMIS 10 Global Physical Health Score
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) 10 - Global Physical Health short form will be administered to all patients to assess their perception of physical health at 12 months. The scale includes a list of questions that patients rate from 1 (poor) which is a minimum value on the scale to 5 (excellent) which is the maximum value on the scale. A higher score indicates a better quality of life.
  The raw scores from the questions are converted into standardized t-scores. In the U.S. general population, the t-score has a mean of 50 and a standard deviation of 10. A t-score higher than 50 indicates a better quality of life compared to the general population. The cut points for the t-score are as follows: above 58 (excellent), 50 to 58 (very good), 42 to 50 (good), 35 to 42 (fair), below 35 (poor).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
T-score | 51.58 (8.30) | 46.60 (8.24)

7. Secondary Outcome: Subclinical Atherosclerosis - IMT
Description: This will be assessed through measures of carotid intima-media thickness (IMT)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
millimeters | 0.58 (0.12) | 0.57 (0.12)

8. Secondary Outcome: Functional Capacity - Strength (Away)
Description: This will be assessed through measures of unilateral isometric strength utilizing Biodex. This measurement is for Away Peak 75-Peak Strength
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
Pounds | 108.02 (48.15) | 100.01 (32.44)

9. Secondary Outcome: Regular Physical Activity Using Accelerometers
Description: Physical activity is assessed through accelerometers which give scores that are measured in m/s^2
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: m/s^2
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
m/s^2 | 16.46 (13.54) | 11.75 (9.17)

10. Secondary Outcome: Metabolic State and Kidney Function - Serum Creatinine (SCr)
Description: Serum creatinine levels will be measured.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
mg/dL | 1.46 (0.50) | 1.37 (0.80)

11. Secondary Outcome: Quality of Life and Perceived Health Status - PROMIS 29 Physical Function Score
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) 29 form will be administered to all patients to assess their perception of their physical function12 months. The scale includes a list of questions that patients rate from 1 (poor) which is a minimum value on the scale to 5 (excellent) which is the maximum value on the scale. A higher score indicates a better quality of life.
  The raw scores from the questions are converted into standardized t-scores. In the U.S. general population, the t-score has a mean of 50 and a standard deviation of 10. A t-score higher than 50 indicates a better quality of life compared to the general population. The cut points for the t-score are as follows: above 45 (within normal limits), 45 to 40 (mild), 30 to 40 (moderate), below 30 (severe).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
T-score | 48.89 (8.64) | 46.45 (10.12)

12. Secondary Outcome: Quality of Life and Perceived Health Status - PROMIS 10 Global Mental Health Score
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) 10 - Global Mental Health short form will be administered to all patients to assess their perception of their mental health at 12 months. The scale includes a list of questions that patients rate from 1 (poor) which is a minimum value on the scale to 5 (excellent) which is the maximum value on the scale. A higher score indicates a better quality of life.
  The raw scores from the questions are converted into standardized t-scores. In the U.S. general population, the t-score has a mean of 50 and a standard deviation of 10. A t-score higher than 50 indicates a better quality of life compared to the general population. The cut points for the t-score are as follows: above 56 (excellent), 48 to 56 (very good), 40 to 48 (good), 29 to 40 (fair), below 29 (poor).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
T-score | 53.11 (7.95) | 49.53 (6.69)

13. Secondary Outcome: Functional Capacity - Strength (Towards)
Description: This will be assessed through measures of unilateral isometric strength utilizing Biodex. This measurement is for Towards Peak 75-Peak Strength
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
Pounds | 44.53 (19.3) | 41.61 (17.62)

14. Secondary Outcome: Pain Intensity
Description: Pain intensity is measured using PROMIS 29 scale. The scale includes a pain intensity question that patients rate from 1 (no pain) to 10 (extreme pain). A higher score indicates higher pain level.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
units on a scale | 1.98 (2.59) | 3.21 (3.02)

15. Secondary Outcome: Body Composition - Waist Circumference
Description: Waist circumference will be measured at the narrowest part of the torso (above the umbilicus and below xiphoid process) in the standing position using a tape measure
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
Inches | 45.50 (7.33) | 45.33 (9.01)

16. Secondary Outcome: Body Composition - Body Mass Index (BMI)
Description: Body mass index is calculated as weight (kg) divided by height (m) squared
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
kg/m^2 | 35.90 (8.12) | 35.12 (10.03)

17. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure will be measured in the supine position (lying on back) in a dimly lit room after resting for fifteen minutes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
mmHg | 132.92 (15.69) | 129.71 (17.22)

18. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 17
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise Rehabiliation | Control
Number analyzed (Participants) | 52 | 28
mmHg | 80.83 (10.71) | 82.46 (9.12)

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed in this study due to the minimal risk associated with the exercise program.
Description: There are minimal to no risks associated with the exercise program.
Arm/Group | Exercise Rehabiliation | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT02409901/Prot_SAP_000.pdf